CLINICAL TRIAL: NCT01382199
Title: A Phase III Randomized, Double Blind, Placebo Controlled, Multicenter Study to Evaluate the Efficacy and Safety of Recombinant Human Lactoferrin Administered Orally for the Prevention of Antibiotic Associated Diarrhea in Adult Patients
Brief Title: Recombinant Human Lactoferrin Administered Orally for the Prevention of Antibiotic Associated Diarrhea in Adult Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ventria Bioscience (Industry)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Dr. Ning Huang, Vice President Research & Development, Ventria Bioscience
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: VB-Ven100-2011-01; R44AG037211 (NIH)
Record Dates: First submitted 2011-06-21; First posted 2011-06-27 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Diarrhea
Keywords: Antibiotic Associated Diarrhea in Adult Patients
MeSH Terms: conditions — Diarrhea | interventions — Lactoferrin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ven100 (Experimental): Recombinant Human Lactoferrin Administered Orally for the Prevention of Antibiotic Associated Diarrhea in Adult Patients
  Interventions: Drug: Lactoferrin

INTERVENTIONS:
Drug: Lactoferrin

SUMMARY:
The purpose of the study is to Evaluate the Efficacy and Safety of Recombinant Human Lactoferrin Administered Orally for the Prevention of Antibiotic Associated Diarrhea in Adult Patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients must meet all of the inclusion criteria listed below at the time of enrollment.

  1. Male and female patients 50 years of age and older.
  2. Resident of a participating long term care facility.
  3. Able to consume 30 mL of liquid solution two time per day by mouth or enteral feeding tube.
  4. Patient has had no antibiotics in the 4 weeks preceding enrollment in the study.
  5. Patient has been started on a broad spectrum antibiotic(s) for an infection other than gastroenteritis.
  6. Patient has a life expectancy greater than 6 months.
  7. Patient or health care agent is able and willing to sign a written informed consent.
  8. Patient or caregiver is able and willing to complete diary of daily bowel movement information (number, formed or unformed, time) during any portion of the 8 week study.

Exclusion Criteria:

1. Patient has an ileostomy.
2. Patient has a prior history of major gastrointestinal surgery such as partial small bowel or colon resection or gastric bypass.
3. Patient has a history of inflammatory bowel disease.
4. Patient has a history of chronic diarrhea associated with irritable bowel syndrome or other etiologies.
5. Patient has a history of severe constipation requiring use of enemas or disimpaction within 30 days prior to enrollment.
6. Patient has signs or symptoms of C. difficile infection including diarrhea.
7. Patient has signs or symptoms of acute or chronic diarrhea.
8. Patient has known sensitivity or allergy to rice or rice products.
9. Patient has significant medical problems which in the judgment of the principal investigator or medical monitor may interfere with participation in the study.
10. Patient is not receiving an antibiotic regimen consisting of a broad spectrum antibiotic.
11. Patient has participated in an investigational study using an investigational product within 30 days of randomization.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2011-09; Primary Completion 2013-09 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Reduction in the number of days of antibiotic associated diarrhea during the treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Ning Huang, Ph.D., Study Director — Ventria Bioscience